CLINICAL TRIAL: NCT06089902
Title: EUROAAOCA Registry
Brief Title: European Prospective Registry on Anomalous Aortic Origin of the Coronary Arteries
Acronym: EUROAAOCA
Status: Recruiting | Type: Observational
Sponsor: University of Padova (Other)
Collaborators: IRCCS Policlinico S. Donato (Other); Mitera Children's Hospital, Athens Heart Surgery Institute, Greece (Unknown); Ospedale Civile Ca' Foncello (Other); University Hospital, Ghent (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Azienda Ospedaliera Universitaria Integrata Verona (Other); University Medical Center Groningen (Other); Hospital Universitario La Paz (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); Insel Gruppe AG, University Hospital Bern (Other); Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, PADALINO MASSIMO, Associate Professor, University of Padova
Other Study IDs: EUROAAOCA group
Record Dates: First submitted 2023-10-03; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Congenital Heart Disease; Coronary Artery Anomaly; Sudden Cardiac Death; Surgical Procedure, Unspecified; Diagnosis; Arrhythmia; Heart Defects, Congenital; Adult Children
Keywords: anomalous; coronary; sudden cardiac death
MeSH Terms: conditions — Heart Defects, Congenital; Death, Sudden, Cardiac; Disease; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adult > 30 years: All adult patient > 30 yrs undergoing diagnosis (incidental or not) of anomalous aortic origin of coronary arteries
  Interventions: Procedure: unroofing or other surgery if needed
- Juvenile < 30 yrs: All young patient <30 yrs undergoing diagnosis (incidental or not) of anomalous aortic origin of coronary arteries
  Interventions: Procedure: unroofing or other surgery if needed

INTERVENTIONS:
Procedure: unroofing or other surgery if needed — unroofing of coronary artery
  Other Names: clinical follow up

SUMMARY:
Anomalous aortic origin of a coronary artery (AAOCA) is a group of rare congenital heart defects with various clinical presentations. The lifetime-risk of an individual living with AAOCA is unknown, and data from multicentre registries are urgently needed to adapt current recommendations and guide optimal patient management. The European Registry for AAOCA (EURO-AAOCA) aims to assess differences with regard to AAOCA management between centres.

DETAILED DESCRIPTION:
EURO AAOCA study database on management for "ANOMALOUS AORTIC ORIGIN OF CORONARY ARTERIES.

This is a simple Excel database in 8 sections (see below). The patient's identification (ID) should be anonymous, and can be decided by each center; the investigators suggest to enclose Centre ID number (which is communicated by the leading center) and a sequential number or date of birth (dd/mm/yy).

If no procedure has been done for the patients , it is required to the "PERIPROCEDURAL, SURGICAL DETAILS" and "POSTPROCEDURAL" data sheets (which are outlined in RED). In the "PERIPROCEDURAL" sheet, the participants may refer either to the surgical or non surgical procedure.

Baseline and long term clinical evaluation sections must be completed for all patients.

In the database, there are lists of multiple different variables which are summarized in tables enclosed in the section, in which each item corresponds to a number.

EURO AAOCA Study DATABASE sections

1. Baseline demo and anatomy: it includes demographic data, and anatomical details for each patient; basic anatomy and course can be selected scrolling an enclosed list; remaining data are requested as yes/no answer
2. Baseline symptoms and indications: it includes symptoms info and indications to surgical/interventional/clinical follow up for each patient; symptoms can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text; in particular, the participants are required to distinguish between recreational non-competitive sports (2-3/week) and Competitive (>5 times/week), Reason for diagnosis in asymptomatic patient can be selected scrolling a list.
3. Baseline instrumental: it includes all possible diagnostic methodologies used for first diagnosis; the test is considered abnormal when it is gives diagnosis of AAOCA, and in this case , the participants are required to describe the findings as precise as possible. In particular, for non-surgical patients, the participants are required to provide a date of the first time any instrumental test suspected AAOCA. ECG data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text
4. Periprocedural: if the patient has gone to surgical or interventional management, the participants are required to fill this section: data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text
5. Surgical details: for surgical patients only, the participants are required to fill this section; data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text
6. Post procedural: for surgical or interventional patients only, the participants are required to fill this section; data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text
7. Follow up 1: this section must be filled for all patients (surgical/interventional /only medical management) and must be updated every year and sent back to the coordinator every June 15th, so as to check yearly the patients. The Investigators suggest an annual follow up for at least 5 years in a row. Follow up data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text. T
8. Follow up Instrumental diagnosis: this section must be filled for all patients (surgical/interventional /only medical management) and must be updated every year and sent back to the coordinator every June 15th, so as to check yearly the patients. The investigators suggest to do this for at least 5 years in a row. Follow up data can be selected scrolling an enclosed list; remaining data are requested as yes/no answer or text

ELIGIBILITY:
Inclusion Criteria:

* All patients with a diagnosis of AAOCA (either referred to surgery or to medical follow-up )

Exclusion Criteria:

* isolated high-coronary take-off (≥ 5mm above sino-tubular junction), anomalous origin of a circumflex from the right coronary artery, anomalous course with a normal origin, and association to major congenital heart disease (i.e. Tetralogy of Fallot, transposition of the great arteries, anomalous origin of a coronary from the pulmonary artery).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients undergoing incidental or not diagnosis of AAOCA
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Symptoms at diagnosis and after surgery | 5 years
  The study will assess the presence of symptoms (angina, chest pain, distress, sudden cardiac death-SCD, syncope, aborted SCD) at diagnosis, and after eventual surgical repair, to assess incidence of symptoms in patients with this anomaly and effectiveness of surgery in removing symptoms.
Incidence of postoperative adverse events | 5 years
  The study will assess the incidence of operative death and adverse events after surgery (in those who undergo surgery).
Incidence of adverse events at follow up | 5 years
  The study will assess the incidence of death and adverse events at clinical follow up either in patients who required a surgical repair or in those who did not undergo surgery because of lack of indications.

SECONDARY OUTCOMES:
Incidence of any arrhythmias at Follow up | 5 years
  The study will assess the incidence of any (mostly ventricular) arrhythmias in all patients, either surgical or non surgical
Rate of return to unrestricted competitive sport | 5 years
  The study will assess the rate of return to unrestricted sport and competitive sport activity in all patients, either surgical or non surgical

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Padalino, MD PhD, Principal Investigator — University of Padova
Locations (2):
- Massimo Padalino, Padua, PD, Italy
- Christopher Grani, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No
The anonymized demographic and clinical data underlying this study can be shared on reasonable request to the principal investigator

REFERENCES:
- [Result] Padalino MA, Jegatheeswaran A, Blitzer D, Ricciardi G, Guariento A. Surgery for Anomalous Aortic Origin of Coronary Arteries: Technical Safeguards and Pitfalls. Front Cardiovasc Med. 2021 May 12;8:626108. doi: 10.3389/fcvm.2021.626108. eCollection 2021. PMID 34055925
- [Result] Bigler MR, Kadner A, Raber L, Ashraf A, Windecker S, Siepe M, Padalino MA, Grani C. Therapeutic Management of Anomalous Coronary Arteries Originating From the Opposite Sinus of Valsalva: Current Evidence, Proposed Approach, and the Unknowing. J Am Heart Assoc. 2022 Oct 18;11(20):e027098. doi: 10.1161/JAHA.122.027098. Epub 2022 Oct 7. PMID 36205254
- [Result] Ponzoni M, Frigo AC, Padalino MA. Surgery for Anomalous Aortic Origin of a Coronary Artery (AAOCA) in Children and Adolescents: A Meta-Analysis. World J Pediatr Congenit Heart Surg. 2022 Jul;13(4):485-494. doi: 10.1177/21501351221095424. PMID 35757950
- [Result] Grani C, Padalino MA. Editorial: Coronary Artery Anomalies: A 2020 Review. Front Cardiovasc Med. 2022 Feb 10;9:776951. doi: 10.3389/fcvm.2022.776951. eCollection 2022. No abstract available. PMID 35224033
- [Result] Thiene G, Frescura C, Padalino M, Basso C, Rizzo S. Coronary Arteries: Normal Anatomy With Historical Notes and Embryology of Main Stems. Front Cardiovasc Med. 2021 May 31;8:649855. doi: 10.3389/fcvm.2021.649855. eCollection 2021. PMID 34136540
- [Result] Padalino MA, Franchetti N, Hazekamp M, Sojak V, Carrel T, Frigiola A, Lo Rito M, Horer J, Roussin R, Cleuziou J, Meyns B, Fragata J, Telles H, Polimenakos AC, Francois K, Veshti A, Salminen J, Rocafort AG, Nosal M, Vedovelli L, Guariento A, Vida VL, Sarris GE, Boccuzzo G, Stellin G. Surgery for anomalous aortic origin of coronary arteries: a multicentre study from the European Congenital Heart Surgeons Associationdagger. Eur J Cardiothorac Surg. 2019 Oct 1;56(4):696-703. doi: 10.1093/ejcts/ezz080. PMID 30897195